CLINICAL TRIAL: NCT05732259
Title: Comparative Effect Of Percussive Therapy Device And Manual Myofascial Release Technique To Improve Hamstrings Flexibility In Traffic Wardens
Brief Title: Comparative Effect Of Percussive Therapy Device And Manual Myofascial Release Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zaidmughal001
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Hamstring Sprain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percussion therapy group (Active Comparator): Group A was given Conventional treatment along with percussion therapy with Theragun PRO (1750-2400 rpm).
  •Participants lying in prone position on the couch received percussion therapy with Theragun PRO using standard ball head at speed of 1750 rpm, for total of 90 seconds, split into 3 sets of 30 seconds with 10 seconds rest
  Interventions: Other: Percussion therapy
- Manual Myofascial Release technique group (Active Comparator): Group B was given Conventional treatment along with manual myofascial release technique for 90 sec continuous.
  Interventions: Other: Manual Myofascial Release technique

INTERVENTIONS:
Other: Percussion therapy — Participant lying in prone position on the couch will receive percussion therapy with Theragun PRO using standard ball head at speed of 1750 rpm, for total of 90 seconds, split into 3 sets of 30 seconds with 10 seconds rest.
  Arms: Percussion therapy group
Other: Manual Myofascial Release technique — Manual myofascial release technique for 90 sec continuous.
  Arms: Manual Myofascial Release technique group

SUMMARY:
The present study was concerned with the comparison of effect of Theragun PRO and manual myofascial release technique to improve Hamstrings Flexibility in healthy Adults. It was randomized clinical trial on two groups one got percussion therapy by theragun PRO and other got treatment through manual myofascial release technique. The outcome measure was hamstring flexibility.

DETAILED DESCRIPTION:
Muscular flexibility is an important aspect of normal human function. Limited flexibility has been shown to predispose a person to reduce quality of life. Several studies developed protocols to improve flexibility of muscles, including manual myofascial release techniques, Stretching techniques or Percussive therapy. The studies about the effects of fascia relaxation and stretching techniques on flexibility reported that fascia relaxation increased flexibility of hamstrings. Many treatments likely combines the elements of a conventional massage and vibration therapy.

There is a lack of scientific evidence as to how and if percussive massage treatment affects ROM and muscle strength. To date, there are many studies on effect of percussive therapy on different muscle group, but investigators did not find work on hamstring muscle group. Therefore, it is aimed to find Comparative effect of Percussive therapy device and manual myofascial release technique to improve Hamstrings Flexibility in healthy Adults.

This was a Randomized clinical trial. Sample was taken through simple random sampling. Investigators will perform randomized clinical trial on two groups one got percussion therapy by theragun PRO and other got treatment through manual myofascial release technique. The outcome measure was hamstring flexibility.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years
* Male gender
* Traffic wardens with 5 years field experience
* Participants labeled by Orthopedic surgeon/Physician with reduced flexibility of hamstring muscle group (Unilateral or Bilateral)

Exclusion Criteria:

* Any history of Low back pain.
* Any traumatic History of lower extremity.
* Arthritis
* Sprain or Strain

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-24 (Actual)

PRIMARY OUTCOMES:
Sit to Reach Test (Change is being assessed) | Change from Baseline range of motion at day 4
  A yardstick is placed on the floor and tape is placed across it at a right angle to the 15 inches mark. The client/patient sits with the yardstick between the legs, with the legs extended at right angles to the taped line on the floor. Heels of the feet should touch the edge of the taped line and be about 10 to 12 inches apart.
  The score is the most distant point (cm or in) reached with the fingertips.
Active knee extension test (Change is being assessed) | Change from Baseline range of motion at day 4
  The subject is positioned on the examination table in supine, the lower limb that is'nt examined is positioned in stabilised on the support surface. The opposite limb is elevated so that the hip is in 90degrees of flexion and the knees are extended to reach a position perpendicular to the ground. A lag of 20degrees is considered normal from full extension, anything less than 20degrees is considered as hamstrings tightness. This range needs to be measure using a goniometer placed at the knee with the fulcrum at the lateral epicondyle, the stationary arm parallel to the thigh pointing to the greater trochanter and the moveable arm parallel to the leg pointing to the lateral malleoli.

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Mughal, DPT, Principal Investigator — University of Lahore
Locations (1):
- Sehat Medical Complex, Lahore, Lahore, Punjab Province, Pakistan